CLINICAL TRIAL: NCT04361500
Title: Registry for the Evaluation of Safety and Effectiveness of the Seraph 100 Microbind Affinity Blood Filter in the Therapy of COVID-19 Patients (COSA)
Brief Title: Registry of COVID-19 Patients Treated With the Seraph 100 Microbind Affinity Blood Filter
Acronym: COSA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Collaborators: Medical Clinic V Nephrology, Academic Teaching Hospital Brunswick (Unknown)
Responsible Party: Sponsor
Other Study IDs: COSA-8998
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- COVID-19 patients with Seraph 100 therapy
  Interventions: Device: Seraph 100

INTERVENTIONS:
Device: Seraph 100 — Seraph 100 therapy during a COVID-19 infection

SUMMARY:
The purpose of this registry study is to investigate the effectiveness and safety of the Seraph® 100 Microbind® Affinity Blood Filter (Seraph 100) in the treatment of COVID-19 patients.

DETAILED DESCRIPTION:
During the ongoing COVID-19 pandemic, millions of people have been infected with SARS- Cov-2 worldwide. In the absence of an approved vaccine or medical treatment, there is an emerging need for treatment options, especially in critically ill patients. Multiple pharmacological and non-pharmacological therapies are being investigated. In 2019, the Seraph® 100 Microbind® Affinity Blood Filter (ExThera Medical Corporation, CA, USA) was approved for the removal of pathogens in Europe. On April 17th the FDA granted Authorization for Emergency Use in patients with COVID-19 admitted to the ICU with confirmed or imminent respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 infection
* Treatment with the Seraph® 100 Microbind® Affinity Blood Filter
* Voluntary consent to participate in Registry

Exclusion Criteria:

- none

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with prooven COVID-19 infection with confirmed or imminent respiratory failure and Treatment with the Seraph® 100 Microbind® Affinity Blood Filter.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Survival | 30 days
  Overall Survival after Seraph 100 therapy session

SECONDARY OUTCOMES:
Length of ICU stay | 30 days
  Time spend in the ICU after Seraph 100 therapy session
Length of Hospital stay | 30 days
  Time spend in the hospital after Seraph 100 therapy session
Length of ventilator therapy | 30 days
  Time spend on ventilator after Seraph 100 therapy session
Adverse events | 30 days
  Report of any Seraph 100 therapy related adverse events

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Academic Teaching Hospital Brunswick, Braunschweig, Lower Saxony
  - Hannover Medical School, Hanover

IPD SHARING:
Plan to Share IPD: No